CLINICAL TRIAL: NCT03074526
Title: Prospective, Double Blinded Randomized Multi-Center Controlled Trial Evaluating the 2 Different Doses of Lyophilized Amniotic Fluid Compared to a Saline Placebo Injection in the Treatment of Subjects With Osteoarthritic (OA) Knee Pain
Brief Title: Protocol for the Clinical Evaluation of Lyophilized Amniotic Fluid in the Treatment of Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OFORT003
Record Dates: First submitted 2017-01-27; First posted 2017-03-08 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Approximately 180 subjects will be enrolled in one of three dose arms ( 4ml, Saline Placebo and 4ml 2x).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 4mL amniotic fluid (Active Comparator): Amniotic Fluid: 4mL dose of amniotic fluid
  Interventions: Other: Amniotic Fluid
- 4mL2x amniotic fluid (Active Comparator): Amniotic Fluid: 4mL 2x dose of amniotic fluid
  Interventions: Other: Amniotic Fluid
- 4mL Saline Placebo (Placebo Comparator): Normal Saline
  Interventions: Other: Saline Placebo

INTERVENTIONS:
Other: Amniotic Fluid — Amniotic Fluid
  Arms: 4mL amniotic fluid; 4mL2x amniotic fluid
Other: Saline Placebo — Saline Placebo
  Arms: 4mL Saline Placebo

SUMMARY:
To evaluate the efficacy of Lyophilized amniotic fluid as compared to the Saline Injection, placebo control in the treatment of moderate osteoarthritis of the knee.

DETAILED DESCRIPTION:
Approximately 180 subjects will be enrolled in one of three dose arms ( 4ml, Saline Placebo and 4ml 2x). The estimated enrollment period is 6 months. Each subject will receive 1 injection and be evaluated for efficacy and safety during a 6 month observation period. The study is expected to be completed within 12 months, inclusive of enrollment and follow-up for all subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 30 years or older.
2. Subject has a diagnosis of osteoarthritis (OA) defined as Grade 1 to 3 on the Kellgren Lawrence grading scale.
3. Subject is willing and able provide informed consent and participate in all procedures and follow-up evaluations necessary to complete the study.
4. Subject must have a VAS pain scale greater than 30.

Exclusion Criteria:

1. Subject has active infection at the injection site.
2. Subject has rheumatoid arthritis, psoriatic arthritis, or have been diagnosed with any other auto-immune disorders that could be the cause of their knee pain.
3. BMI greater than 45 kg/m2
4. Subject has received an intra-articular hyaluronic acid (HA) injection for the treatment of OA of the target knee within 12 weeks prior to screening.
5. Subject has received a steroid or platelet rich plasma (PRP) injection for the treatment of OA of the target knee within 12 weeks prior to screening.
6. Subject has had major surgery or arthroscopy in the target knee within 26 weeks of treatment or plans to have surgery in the target knee within 180 days of treatment.
7. Subject is pregnant or plans to become pregnant within 180 days of treatment.
8. Subject has used an investigational drug, device or biologic within 12 weeks prior to treatment.
9. Subject has any significant medical condition that, in the opinion of the Investigator, would interfere with protocol evaluation and participation.
10. Subject has a history of immunosuppressive or chemotherapy in the last 5 years
11. Subject has autoimmune disease or a known history of having Acquired Immunodeficiency Syndromes (AIDS) or HIV
12. Subject has had prior radiation at the site
13. Subject is currently taking anticoagulant therapy (excluding Plavix or Aspirin)
14. New diagnosis of gout in the past 6 month
15. Subject has a diagnosis of osteoarthritis (OA) defined as Grade 4 on the Kellgren Lawrence grading scale.
16. Subject has a diagnosis of Osteonecrosis of the knee.
17. Subject has had a total knee replacement.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2018-04-25 (Actual)

PRIMARY OUTCOMES:
Reduction in Pain | 3 month
  The proportion of subjects who experience at least 20% improvement over baseline in Visual Analog Scale for Pain at 3 months in the Lyophilized amniotic fluid Injectable versus placebo-treated group.

SECONDARY OUTCOMES:
Range of Motion | 3 months
  subjects who experience a level of improvement in function as assessed by range of motion at 3 months
Knee Injury and Osteoarthritis Outcome Score | 4weeks, 6weeks, 3 months, 16 weeks, 6 months
  measurement to assess the patient's opinion about their knee and associated problems by looking at pain, functions of daily living, function in sports and recreation, knee related quality of life and other symptoms
SF-12 Health Health Survey | 4weeks, 6weeks, 3 months, 16 weeks, 6 months
  patient-reported survey assessing patient health
Activity of Daily Living Questionnaire | 4weeks, 6weeks, 3 months, 16 weeks, 6 months
  Changes in the subject's physical activity level

CONTACTS AND LOCATIONS:
Overall Officials: David Mason, MD, Study Director — Chief Medical Officer
Locations (4):
- United States (4):
  - Central Research Associates, Inc, Birmingham, Alabama
  - Southeastern Center for Clinical Trials, Atlanta, Georgia
  - Weil Foot, Ankle and Orthopedic Institute, Des Plaines, Illinois
  - Hinsdale Orthopaedic Associates, Hinsdale, Illinois

IPD SHARING:
Plan to Share IPD: No